CLINICAL TRIAL: NCT02279277
Title: Effect of Physical Therapy on Grade 3 or 4 Knee Osteoarthritis
Brief Title: Physical Therapy Prior to Total Knee Replacement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Austin2014
Record Dates: First submitted 2014-10-06; First posted 2014-10-31 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-10

CONDITIONS: Osteoarthritis of the Hip
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No physical therapy (No Intervention): No prescribed, supervised physical therapy prior to total knee replacement
- Physical Therapy (Active Comparator): Prescribed, supervised physical therapy prior to total knee replacement
  Interventions: Behavioral: Supervised physical therapy program prior to total knee replacement surgery

INTERVENTIONS:
Behavioral: Supervised physical therapy program prior to total knee replacement surgery
  Arms: Physical Therapy

SUMMARY:
In this study, the investigators are investigating the effects of physical therapy (PT) for treating high grade knee osteoarthritis (OA) in patients that are candidates for total knee replacement. Through the examination of patient outcomes, such as pain, stiffness, and physical function, the investigators will determine if PT prior to total knee replacement is an effective treatment in a patient with high grade OA.

ELIGIBILITY:
Inclusion Criteria:

1. Knee osteoarthritis (Kellgren-Lawrence grade 3 or 4) confirmed via standing AP radiograph
2. Surgical candidate for TKA, having had a least a 3 months of pain affecting ADL's unresponsive to conservative treatment consisting of AT LEAST one non-narcotic medication AND one injection (corticosteroid or series of viscosupplementation). Injection must not have been administered within 6 weeks of start of PT trial
3. Prior knee surgery from arthroscopies, meniscal surgery and ligament reconstruction

Exclusion Criteria:

1. Anyone who received physical therapy in the last 6 months
2. Inability to walk unaided for >1 block
3. Currently engaged in regular PT or a regular home exercise program
4. Prior knee arthroplasty
5. Prior knee surgery for trauma, tumor and osteotomy
6. Injection given within 6 weeks of starting therapy
7. Patients using daily narcotic medications within prior 6 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Range of Motion following Total Knee Replacement | 6 weeks

SECONDARY OUTCOMES:
Patient reported perception of pain following total knee replacement | 6 weeks
Return to functional activities following total knee replacement | 6 weeks